CLINICAL TRIAL: NCT00679679
Title: Clinical Metabolic and Endocrine Parameters in Response to Metformin and Lifestyle Intervention in Women With Polycystic Ovary Syndrome: A Phase 4 Randomized, Double- Blind and Placebo Control Trial
Brief Title: Metformin and Lifestyle Intervention in Women With Polycystic Ovary Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Privado de Cordoba, Argentina (Other)
Responsible Party: Dr. Carolina Fux Otta, Hospital Privado de Córdoba, Argentina
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Fux-1
Record Dates: First submitted 2008-05-15; First posted 2008-05-19 (Estimated); Last update posted 2008-05-19 (Estimated); Status verified 2008-05

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Polycystic ovary syndrome; Treatment; Metformin
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metformin (Experimental): Every patient will be given diet and exercise counseling in both arms. Intervention arm will receive metformin
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator): Every patient will be given diet and exercise counseling in both arms. Intervention arm will receive metformin
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — Metformin 750 mg BID for 4 months
  Other Names: D.B.I. 500 mg. 1 1/2 tables BID
  Arms: Metformin
Drug: Placebo — Diet counseling and exercise
  Arms: Placebo

SUMMARY:
Polycystic ovary syndrome is a frequent cause of abnormal menses and infertility. It has also been related to cardiovascular disease.

The objective of this trial is to evaluate the clinical and metabolic efficacy of metformin plus life style modifications in women with polycystic ovary syndrome compared with life style modifications and placebo

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is a common and heterogeneous disorder of women in reproductive age. It is characterized by hyperandrogenism and chronic anovulation. Several studies in diverse populations estimate it's prevalence at 5-10%. Women present, in a high percentage of cases, with obesity, hirsutism, acne, menstrual irregularities and infertility. Although the exact physiopathology of PCOS remains unknown, several studies tend to point to insulinoresistance (IR) as the cause of the syndrome. IR is present in 60 to 70% of patients independently of obesity. Compensatory hyperinsulinism has a pivotal role in the physiopathogenesis of PCOS. In vitro, insulin stimulates androgen synthesis in thecal cells and decrease sex hormone-binding globulin synthesis in the liver, increasing free androgen availability.

Due to the high prevalence of IR, PCOS shares components of metabolic syndrome: abdominal obesity, impaired glucose tolerance, gestational and type 2 diabetes, abnormalities in lipid profile, blood hypertension, endothelial dysfunction and probably cardiovascular disease.

In the past, PCOS treatment was focus on ovulation induction for infertility, oral contraceptives for irregular bleeding, and androgens antagonists for hirsutism or acne. In later years insulin sensitizing agents have been used to reduce hyperinsulinemia, improve ovary function and associated metabolic abnormalities. Metformin (MTF), a biguanide, usually used in obese patients with type 2 diabetes,inhibits glucose hepatic production,decreases insulin secretion and increases peripheral insulin sensitivity.

Some studies have reported an improvement in insulin sensitivity associated with reduction of hyperandrogenism and improvements in reproductive abnormalities with MTF. On the other hand, other authors failed to observe those changes. However, an off label indication for it usage in PCOS for FDA and the lack of large controlled trials, MTF indication to treat PCOS has grown dramatically in later years.

In obese women with PCOS, weight loss effectively ameliorates hyperandrogenism and metabolic disorders by improving insulin resistance.

Some trials have suggested that those effects could be improved with insulin sensitizing agents without changes in body weigh.

The present study was designed to assess, in a randomized, double-blind, placebo-controlled way, the effects of MTF in addition to lifestyle modifications on endocrine and metabolic disturbances in women with PCOS.

ELIGIBILITY:
Inclusion Criteria:

* Women in reproductive age
* With polycystic ovary syndrome defined by hyperandrogenism (elevated serum testosterone concentrations), and oligomenorrhea (cycles of 35 days or longer), or amenorrhea (no menses in the last 6 months) after negative screening pregnancy test

Exclusion Criteria:

* Pregnancy
* Cushing' s syndrome
* Late onset congenital adrenal hyperplasia
* Androgen-secreting tumors
* Uncontrolled thyroid disease
* Hyperprolactinemia
* Diabetes any
* Cardiovascular diseases (Ischaemic heart disease, uncontrolled hypertension, heart failure)
* Acute or chronic infections at baseline
* Renal disease
* Liver disease
* Had taken any medications for at least 3 months before enrolment in the study.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2003-01; Primary Completion 2005-09 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Body mass index,Normalization of menses,Pregnancy,Hirsutism,Waist to hip ratio, Testosterone, Androstenedione, DHEAS,Progesterone, FSH, LH,Glucose, OGTT,Insulinemia,Total HDL and LDL Cholesterol, Triglycerides,Uric acid, Prostate specific antigen | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Carolina Fux Otta, MD, Principal Investigator
Locations (1):
- Hospital Privado de Córdoba, Córdoba, Córdoba Province, Argentina

REFERENCES:
- [Background] Azziz R, Woods KS, Reyna R, Key TJ, Knochenhauer ES, Yildiz BO. The prevalence and features of the polycystic ovary syndrome in an unselected population. J Clin Endocrinol Metab. 2004 Jun;89(6):2745-9. doi: 10.1210/jc.2003-032046. PMID 15181052
- [Background] Asuncion M, Calvo RM, San Millan JL, Sancho J, Avila S, Escobar-Morreale HF. A prospective study of the prevalence of the polycystic ovary syndrome in unselected Caucasian women from Spain. J Clin Endocrinol Metab. 2000 Jul;85(7):2434-8. doi: 10.1210/jcem.85.7.6682. PMID 10902790
- [Background] Diamanti-Kandarakis E, Kouli CR, Bergiele AT, Filandra FA, Tsianateli TC, Spina GG, Zapanti ED, Bartzis MI. A survey of the polycystic ovary syndrome in the Greek island of Lesbos: hormonal and metabolic profile. J Clin Endocrinol Metab. 1999 Nov;84(11):4006-11. doi: 10.1210/jcem.84.11.6148. PMID 10566641
- [Background] Ehrmann DA. Polycystic ovary syndrome. N Engl J Med. 2005 Mar 24;352(12):1223-36. doi: 10.1056/NEJMra041536. No abstract available. PMID 15788499
- [Background] Dunaif A. Insulin resistance and the polycystic ovary syndrome: mechanism and implications for pathogenesis. Endocr Rev. 1997 Dec;18(6):774-800. doi: 10.1210/edrv.18.6.0318. PMID 9408743
- [Background] Dunaif A, Segal KR, Futterweit W, Dobrjansky A. Profound peripheral insulin resistance, independent of obesity, in polycystic ovary syndrome. Diabetes. 1989 Sep;38(9):1165-74. doi: 10.2337/diab.38.9.1165. PMID 2670645
- [Background] Barbieri RL, Makris A, Randall RW, Daniels G, Kistner RW, Ryan KJ. Insulin stimulates androgen accumulation in incubations of ovarian stroma obtained from women with hyperandrogenism. J Clin Endocrinol Metab. 1986 May;62(5):904-10. doi: 10.1210/jcem-62-5-904. PMID 3514651
- [Background] Nestler JE, Powers LP, Matt DW, Steingold KA, Plymate SR, Rittmaster RS, Clore JN, Blackard WG. A direct effect of hyperinsulinemia on serum sex hormone-binding globulin levels in obese women with the polycystic ovary syndrome. J Clin Endocrinol Metab. 1991 Jan;72(1):83-9. doi: 10.1210/jcem-72-1-83. PMID 1898744
- [Background] Alberti KG, Zimmet P, Shaw J; IDF Epidemiology Task Force Consensus Group. The metabolic syndrome--a new worldwide definition. Lancet. 2005 Sep 24-30;366(9491):1059-62. doi: 10.1016/S0140-6736(05)67402-8. No abstract available. PMID 16182882
- [Background] Legro RS, Kunselman AR, Dodson WC, Dunaif A. Prevalence and predictors of risk for type 2 diabetes mellitus and impaired glucose tolerance in polycystic ovary syndrome: a prospective, controlled study in 254 affected women. J Clin Endocrinol Metab. 1999 Jan;84(1):165-9. doi: 10.1210/jcem.84.1.5393. PMID 9920077
- [Background] Christian RC, Dumesic DA, Behrenbeck T, Oberg AL, Sheedy PF 2nd, Fitzpatrick LA. Prevalence and predictors of coronary artery calcification in women with polycystic ovary syndrome. J Clin Endocrinol Metab. 2003 Jun;88(6):2562-8. doi: 10.1210/jc.2003-030334. PMID 12788855
- [Background] Wild RA. Long-term health consequences of PCOS. Hum Reprod Update. 2002 May-Jun;8(3):231-41. doi: 10.1093/humupd/8.3.231. PMID 12078834
- [Background] Dahlgren E, Janson PO, Johansson S, Lapidus L, Oden A. Polycystic ovary syndrome and risk for myocardial infarction. Evaluated from a risk factor model based on a prospective population study of women. Acta Obstet Gynecol Scand. 1992 Dec;71(8):599-604. doi: 10.3109/00016349209006227. PMID 1336918
- [Background] Talbott E, Clerici A, Berga SL, Kuller L, Guzick D, Detre K, Daniels T, Engberg RA. Adverse lipid and coronary heart disease risk profiles in young women with polycystic ovary syndrome: results of a case-control study. J Clin Epidemiol. 1998 May;51(5):415-22. doi: 10.1016/s0895-4356(98)00010-9. PMID 9619969
- [Background] Paradisi G, Steinberg HO, Hempfling A, Cronin J, Hook G, Shepard MK, Baron AD. Polycystic ovary syndrome is associated with endothelial dysfunction. Circulation. 2001 Mar 13;103(10):1410-5. doi: 10.1161/01.cir.103.10.1410. PMID 11245645
- [Background] Sam S, Dunaif A. Polycystic ovary syndrome: syndrome XX? Trends Endocrinol Metab. 2003 Oct;14(8):365-70. doi: 10.1016/j.tem.2003.08.002. PMID 14516934
- [Background] Matthaei S, Stumvoll M, Kellerer M, Haring HU. Pathophysiology and pharmacological treatment of insulin resistance. Endocr Rev. 2000 Dec;21(6):585-618. doi: 10.1210/edrv.21.6.0413. PMID 11133066
- [Background] Harborne L, Fleming R, Lyall H, Norman J, Sattar N. Descriptive review of the evidence for the use of metformin in polycystic ovary syndrome. Lancet. 2003 May 31;361(9372):1894-901. doi: 10.1016/S0140-6736(03)13493-9. PMID 12788588
- [Background] Norman RJ, Homan G, Moran L, Noakes M. Lifestyle choices, diet, and insulin sensitizers in polycystic ovary syndrome. Endocrine. 2006 Aug;30(1):35-43. doi: 10.1385/ENDO:30:1:35. PMID 17185790
- [Background] Azziz R, Ehrmann D, Legro RS, Whitcomb RW, Hanley R, Fereshetian AG, O'Keefe M, Ghazzi MN; PCOS/Troglitazone Study Group. Troglitazone improves ovulation and hirsutism in the polycystic ovary syndrome: a multicenter, double blind, placebo-controlled trial. J Clin Endocrinol Metab. 2001 Apr;86(4):1626-32. doi: 10.1210/jcem.86.4.7375. PMID 11297595
- [Background] Velazquez EM, Mendoza S, Hamer T, Sosa F, Glueck CJ. Metformin therapy in polycystic ovary syndrome reduces hyperinsulinemia, insulin resistance, hyperandrogenemia, and systolic blood pressure, while facilitating normal menses and pregnancy. Metabolism. 1994 May;43(5):647-54. doi: 10.1016/0026-0495(94)90209-7. PMID 8177055
- [Background] Tepper SL, Jagirdar J, Heath D, Geller SA. Homology between the female paraurethral (Skene's) glands and the prostate. Immunohistochemical demonstration. Arch Pathol Lab Med. 1984 May;108(5):423-5. PMID 6546868
- [Background] Clements J, Mukhtar A. Glandular kallikreins and prostate-specific antigen are expressed in the human endometrium. J Clin Endocrinol Metab. 1994 Jun;78(6):1536-9. doi: 10.1210/jcem.78.6.7515392.
- [Background] Cassidenti DL, Paulson RJ, Serafini P, Stanczyk FZ, Lobo RA. Effects of sex steroids on skin 5 alpha-reductase activity in vitro. Obstet Gynecol. 1991 Jul;78(1):103-7. PMID 1828548
- [Background] Escobar-Morreale HF, Serrano-Gotarredona J, Avila S, Villar-Palasi J, Varela C, Sancho J. The increased circulating prostate-specific antigen concentrations in women with hirsutism do not respond to acute changes in adrenal or ovarian function. J Clin Endocrinol Metab. 1998 Jul;83(7):2580-4. doi: 10.1210/jcem.83.7.4960. PMID 9661648
- [Background] Kuhl H. Comparative pharmacology of newer progestogens. Drugs. 1996 Feb;51(2):188-215. doi: 10.2165/00003495-199651020-00002. PMID 8808163
- [Background] Zarghami N, Grass L, Sauter ER, Diamandis EP. Prostate-specific antigen in serum during the menstrual cycle. Clin Chem. 1997 Oct;43(10):1862-7. PMID 9342005
- [Background] Morin-Papunen L, Vauhkonen I, Koivunen R, Ruokonen A, Martikainen H, Tapanainen JS. Metformin versus ethinyl estradiol-cyproterone acetate in the treatment of nonobese women with polycystic ovary syndrome: a randomized study. J Clin Endocrinol Metab. 2003 Jan;88(1):148-56. doi: 10.1210/jc.2002-020997. PMID 12519844
- [Background] Lord JM, Flight IH, Norman RJ. Metformin in polycystic ovary syndrome: systematic review and meta-analysis. BMJ. 2003 Oct 25;327(7421):951-3. doi: 10.1136/bmj.327.7421.951. PMID 14576245
- [Background] Lord JM, Flight IH, Norman RJ. Insulin-sensitising drugs (metformin, troglitazone, rosiglitazone, pioglitazone, D-chiro-inositol) for polycystic ovary syndrome. Cochrane Database Syst Rev. 2003;(3):CD003053. doi: 10.1002/14651858.CD003053. PMID 12917943
- [Background] Guzelmeric K, Seker N, Unal O, Turan C. High serum prostate-specific antigen concentrations in hirsute women do not decrease with treatment by the combination of spironolactone and the contraceptive pill. Gynecol Endocrinol. 2004 Oct;19(4):190-5. doi: 10.1080/09513590400012069. PMID 15724801
- [Background] Escobar-Morreale HF, Avila S, Sancho J. Serum prostate-specific antigen concentrations are not useful for monitoring the treatment of hirsutism with oral contraceptive pills. J Clin Endocrinol Metab. 2000 Jul;85(7):2488-92. doi: 10.1210/jcem.85.7.6664. PMID 10902798
- [Background] Bahceci M, Bilge M, Tuzcu A, Tuzcu S, Bahceci S. Serum prostate specific antigen levels in women with polycystic ovary syndrome and the effect of flutamide+desogestrel/ethinyl estradiol combination. J Endocrinol Invest. 2004 Apr;27(4):353-6. doi: 10.1007/BF03351061. PMID 15233555
- [Background] Negri C, Tosi F, Dorizzi R, Fortunato A, Spiazzi GG, Muggeo M, Castello R, Moghetti P. Antiandrogen drugs lower serum prostate-specific antigen (PSA) levels in hirsute subjects: evidence that serum PSA is a marker of androgen action in women. J Clin Endocrinol Metab. 2000 Jan;85(1):81-4. doi: 10.1210/jcem.85.1.6230. PMID 10634368
- [Background] Rosner W, Auchus RJ, Azziz R, Sluss PM, Raff H. Position statement: Utility, limitations, and pitfalls in measuring testosterone: an Endocrine Society position statement. J Clin Endocrinol Metab. 2007 Feb;92(2):405-13. doi: 10.1210/jc.2006-1864. Epub 2006 Nov 7. PMID 17090633
- [Background] Gullu S, Emral R, Asik M, Cesur M, Tonyukuk V. Diagnostic value of prostatic specific antigen in hirsute women. J Endocrinol Invest. 2003 Dec;26(12):1198-202. doi: 10.1007/BF03349157. PMID 15055472
- [Background] Rotterdam ESHRE/ASRM-Sponsored PCOS consensus workshop group. Revised 2003 consensus on diagnostic criteria and long-term health risks related to polycystic ovary syndrome (PCOS). Hum Reprod. 2004 Jan;19(1):41-7. doi: 10.1093/humrep/deh098. PMID 14688154
- [Derived] Fux Otta C, Wior M, Iraci GS, Kaplan R, Torres D, Gaido MI, Wyse EP. Clinical, metabolic, and endocrine parameters in response to metformin and lifestyle intervention in women with polycystic ovary syndrome: a randomized, double-blind, and placebo control trial. Gynecol Endocrinol. 2010 Mar;26(3):173-8. doi: 10.3109/09513590903215581. PMID 20148739